CLINICAL TRIAL: NCT05772546
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of Avatrombopag for Persistent Chemotherapy-Induced Thrombocytopenia in Patients With Gastrointestinal Malignancies (ACT-GI)
Brief Title: Avatrombopag vs. Placebo for CIT in GI Malignancies
Acronym: ACT-GI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hanny Al-Samkari, MD (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor-Investigator, Hanny Al-Samkari, MD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-712
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Cancer; Gastrointestinal Neoplasms; Chemotherapy-Induced Thrombocytopenia
Keywords: Chemotherapy-Induced Thrombocytopenia; CIT; Gastrointestinal Malignancies; Gastrointestinal Cancer; Gastrointestinal Neoplasms; Avatrombopag; Thrombopoietin; Thrombopoietin receptor agonist
MeSH Terms: conditions — Gastrointestinal Neoplasms; Jacobs syndrome | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A - Avatromopag (Experimental): 30 participants will be randomized into a 1:1 fashion and will be stratified based on the number of cytotoxic agents in the patient's chemotherapy regimen. Participants will complete study procedures as outlined:
  Lead-In Period (Day 1 - 15)
  * Pre-determined dose of Avatrombopag 1x daily.
  * Participants failing to achieve a platelet count ≥100,000/µL within 2 weeks will be considered a treatment failure (and will proceed to the end-of-study visit).
  On-Cycle Period (Day 15 - up to Week 6)
  • Pre-determined dose of Avatrombopag 1x daily.
  Follow-up Period
  * End of Treatment on-site visit.
  * Follow-up visit 30-42 days after End of Treatment visit.
  Interventions: Drug: Avatrombopag
- Group B - Matching Placebo (Active Comparator): 30 participants will be randomized into a 1:1 fashion and will be stratified based on the number of cytotoxic agents in the patient's chemotherapy regimen. Participants will complete study procedures as outlined:
  Lead-In Period (Day 1 - 15)
  * Pre-determined dose of matching placebo 1x daily.
  * Participants failing to achieve a platelet count ≥100,000/µL within 2 weeks will be considered a treatment failure (and will proceed to the end-of-study visit).
  On-Cycle Period (Day 15 - up to Week 6)
  • Pre-determined dose of matching placebo 1x daily.
  Follow-up Period
  * End of Treatment on-site visit.
  * Follow-up visit 30-42 days after End of Treatment visit.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Avatrombopag — Thrombopoietin receptor agonist, tablet taken orally.
  Other Names: Doptelet, avatrombopag maleate
  Arms: Group A - Avatromopag
Drug: Matching Placebo — Lactose monohydrate, tablet taken orally.
  Arms: Group B - Matching Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of two study drugs, Avatrobopag versus placebo, to treat persistent Chemotherapy-Induced Thrombocytopenia (CIT) in patients with gastrointestinal (GI) malignancies receiving cytotoxic chemotherapy.

The names of the study drugs involved in this study are:

* Avatrombopag (a thrombopoietin receptor agonist)
* Matching placebo

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, multicenter phase 2 clinical trial evaluating Avatrombopag versus placebo for Chemotherapy-Induced Thrombocytopenia (CIT) in patients with gastrointestinal (GI) malignancies. Avatrombopag may increase or stimulate megakaryocytes, which aid in producing blood platelets, resulting in an increased production of platelets.

* Participants will be "randomized" into one of the study groups: Group A: Avatrombopag or Group B: Matching placebo. Randomization means that a participant is put into a group by chance.
* All patients who complete the study (whether they received avatrombopag or placebo) have the opportunity to receive avatrombopag to treat CIT through a special free drug program available only to the participants of this study.

The U.S. Food and Drug Administration (FDA) has not approved avatrombopag for CIT, but it has been approved for other uses.

Study procedures include screening for eligibility, treatment visits, and blood tests.

Participants will receive the study treatment or placebo for up to seven weeks and will be followed for up to 42 days after the last dose.

It is expected that about 60 people will take part in this research study.

Swedish Orphan Biovitrum (Sobi), biopharmaceutical company, is supporting this research study by providing the study drugs and funding.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of persistent chemotherapy-induced thrombocytopenia, as defined by a platelet count of <85,000/µL on Day 1 of a chemotherapy cycle.
* Age ≥18 years at the time of informed consent. Because no dosing or adverse event data are currently available on the use of avatrombopag for CIT in participants <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Receiving cytotoxic chemotherapy for a gastrointestinal malignancy, including esophageal, gastric, small bowel, hepatobiliary (cholangiocarcinoma, gallbladder carcinoma, hepatocellular carcinoma), pancreatic, or colorectal cancer. Lymphomas are not eligible. Patients of any stage are eligible.
* The chemotherapy regimen being used to treat the patient's gastrointestinal malignancy must be administered in 14, 21, or 28-day cycles and include at least one of the following agents: fluorouracil, capecitabine, floxuridine, trifluridine/tipiracil, gemcitabine, cisplatin, carboplatin, oxaliplatin, irinotecan, liposomal irinotecan, paclitaxel, nanoalbumin-bound paclitaxel, docetaxel, epirubicin, or doxorubicin.
* A plan to continue the current chemotherapy regimen (the regimen that resulted in CIT) at the same dose and schedule for at least 1 more cycle if the platelet count is adequate (>100,000/µL).
* Participant has not received cytotoxic chemotherapy in the 13 days before study Day 1, except for infusional fluorouracil in regimens with a 14-day cycle length or oral cytotoxic chemotherapy agents. .
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (see Appendix B) and a life expectancy of >12 weeks at screening.
* Participants must have adequate organ and marrow function as defined below. Use of standard-of-care G-CSF and/or red cell transfusions to achieve adequate ANC and hemoglobin levels is allowed.

  * Absolute neutrophil count (ANC) ≥500/µL
  * Hemoglobin ≥8 g/dL
  * AST (SGOT) and ALT (SGPT) ≤5 × institutional ULN
  * Total bilirubin ≤3 × institutional ULN
* The effects of avatrombopag on the developing human fetus are unknown. For this reason, women of child-bearing potential and men (except for a vasectomized man with confirmed azoospermia) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for the 30 days after discontinuation of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participant is willing and able to comply with the study protocol.
* Ability to understand and the willingness to sign a written informed consent document, unless the participant lacks capacity to provide consent, in which case a legally authorized representative (LAR) gives permission for the participant to participate.

Exclusion Criteria:

* Participant has a history of hematologic malignancy, including leukemia, lymphoma, myeloma, myelodysplastic syndrome, or a myeloproliferative neoplasm, with the exception of a non-clinically significant neoplasm in the judgement of the investigator (e.g., indolent B-cell neoplasm not requiring treatment, monoclonal gammopathy of undetermined significance, etc.).
* Participant has known bone marrow invasion by tumor or multiple (greater than 1) bony metastatic lesions. Participants do not need to undergo screening with bone marrow biopsy or imaging to satisfy this criterion.
* Participant has received prior irradiation directly to the pelvic bones of a dose of >20 Gy.
* Participants with a history of a prior major venous thromboembolic event, such as a deep vein thrombosis or pulmonary embolism, or symptomatic arterial thrombotic events such as a myocardial infarction, ischemic cerebral vascular accident or transient ischemic attack will be ineligible if they have not tolerated anticoagulation therapy. If patients remain on anticoagulation or have completed the prescribed course of anticoagulation, they will be eligible for enrollment. A venous thrombotic event associated with a central venous catheter or a superficial venous thrombosis will not make the patient ineligible.
* Participant has spontaneous recovery of the platelet count to >100,000/µL prior to randomization.
* Participant has any known clinically significant acute or active bleeding (e.g. gastrointestinal or central nervous system) within 7 days prior to consent.
* Participants who are receiving any other investigational agents or have received any other investigational agent within 30 days of study Day 1.
* History of hypersensitivity reactions to avatrombopag or any of its excipients.
* Participants with uncontrolled intercurrent illness, in the opinion of the investigator.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements, in the opinion of the investigator.
* Pregnant women are excluded from this study because the effect of avatrombopag on the developing fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with avatrombopag, breastfeeding should be discontinued if the mother is treated with avatrombopag. Pregnancy status will be assessed with a serum B-HCG pregnancy test in women of child-bearing potential (see Section 10 for timing). Women who are menopausal or perimenopausal will have follicle-stimulating hormone levels drawn to confirm menopausal status.
* Participant has received a platelet transfusion within 3 days of study Day 1.
* Participant is unable to take oral medication.
* Participant has received a thrombopoietin receptor agonist (romiplostim, eltrombopag, avatrombopag, or lusutrombopag) for any reason within 14 days of study Day 1.
* Participant has a history of active chronic platelet disorders or thrombocytopenia due to an etiology other than CIT, in the opinion of the investigator.
* Any other medical condition or factor that, in the opinion of the investigator, is likely to interfere with completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | Up to 6 weeks
  The primary endpoint of this study is the comparison of the response rate between the avatrombopag arm and the placebo arm. A response is defined as achieving a platelet count ≥100,000/µL within the 2 week lead-in period and then finishing at least 1 cycle of chemotherapy without CIT recurrence (no on-cycle dose-reduction or treatment delay due to thrombocytopenia and ability to receive another cycle of chemotherapy without dose-reduction or treatment delay, defined as platelet count of ≥100,000/µL at the start of the following cycle whether or not an additional cycle is planned).
Response Rate of CIT Treatment in Avatrombopag | Up to 6 weeks
  Defined as the composite of successful initial platelet count recovery to ≥100,000/µL within 15 days of initiation of study drug, plus CIT prevention for one additional chemotherapy cycle (including at the completion of that cycle/start of the following cycle).
Response Rate of CIT Treatment in Placebo Group | Up to 6 weeks
  Defined as the composite of successful initial platelet count recovery to ≥100,000/µL within 15 days of initiation of study drug, plus CIT prevention for one additional chemotherapy cycle (including at the completion of that cycle/start of the following cycle).

SECONDARY OUTCOMES:
Proportion of Platelet Count Recovery in Avatrombopag Group | At baseline, days 8 +/-1 and 15 +/-1
  Assessed by the rate of initial platelet count recovery to ≥100,000/µL during the lead-in period
Proportion of Platelet Count Recovery in Placebo Group | At baseline, days 8 +/-1 and 15 +/-1
  Assessed by the rate of initial platelet count recovery to ≥100,000/µL during the lead-in period.
Requirement of Platelet Transfusions in Avatrombopag Group | Day 1 to 30 days post-treatment discontinuation
  The decision on platelet transfusion could be made either because the patient's platelet count is below a threshold, or due to physician's decision. The probability of patients requiring platelet transfusion will be estimated with a 95% confidence interval.
Requirement of Platelet Transfusions in Placebo Group | Day 1 to 30 days post-treatment discontinuation
  The decision on platelet transfusion could be made either because the patient's platelet count is below a threshold, or due to physician's decision. The probability of patients requiring platelet transfusion will be estimated with a 95% confidence interval.
Rate of Clinically Relevant Bleeding Events in Avatrombopag Group | Day 1 to 30 days post-treatment discontinuation
  The rate of clinically relevant bleeding will be estimated by the Kaplan-Meier curve. Bleeding events will be graded according to CTCAE and according to the modified WHO bleeding scale. Clinically significant bleeding events will be considered grade II-IV events per this scale.
Rate of Clinically Relevant Bleeding Events in Placebo Group | Day 1 to 30 days post-treatment discontinuation
  The rate of clinically relevant bleeding will be estimated by the Kaplan-Meier curve. Bleeding events will be graded according to CTCAE and according to the modified WHO bleeding scale. Clinically significant bleeding events will be considered grade II-IV events per this scale.
Rate of Thromboembolic Events in Avatrombopag Group | Day 1 to 30 days post-treatment discontinuation
  Thromboembolic events will be graded per CTCAE.
Rate of Thromboembolic Events in Placebo Group | Day 1 to 30 days post-treatment discontinuation
  Thromboembolic events will be graded per CTCAE.
Rate of Serious Treatment-Emergent Adverse Events (TEAEs) in Avatromobopag Group | Day 1 to 30 days post-treatment discontinuation
  TEAEs will be graded per CTCAE.
Rate of Serious Treatment-Emergent Adverse Events (TEAEs) in Placebo Group | Day 1 to 30 days post-treatment discontinuation
  TEAEs will be graded per CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Hanny Al-Samkari, MD, Principal Investigator — Massachusetts General Hospital; Gerald A Soff, MD, Principal Investigator — University of Miami Cancer Center
Locations (4):
- United States (4):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Oregon Health and Science University Hospital, Portland, Oregon
  - University of Washington Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation